CLINICAL TRIAL: NCT03676452
Title: The Effects of a Home-based Multicomponent Exergame Training on Motor Functions, Cognition, and Brain Structure of Older Adults: A Multinational Randomized Controlled Trial
Brief Title: The Effects of an Exergame Training on Body and Brain of Older Adults
Acronym: Active@Home
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eling DeBruin (Other)
Responsible Party: Sponsor-Investigator, Eling DeBruin, Professor, Swiss Federal Institute of Technology
Organization: Swiss Federal Institute of Technology (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: BASEC-Nr. 2018-00510
Record Dates: First submitted 2018-08-27; First posted 2018-09-18 (Actual); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Fall Prevention in Healthy Aging

STUDY DESIGN:
Intervention Model Description: This is a two-arm randomized controlled trial with an intervention group and a usual care waitlist control group. After pre-measurement, participants of the intervention group train for four months with the Active@Home exergame. Participants of the control group are instructed to continue their usual daily business and activities. Then, post-measurement takes place. After post-measurement, participants of the control group get the Active@Home exergame for their personal use at home (for several months, no additional measurement).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants of the intervention group train for 16 weeks (three times per week) with a multicomponent virtual reality-based exergame at their home. The Active@Home exergame contains strength training with Tai Chi-based exercises, balance training with dancing and a cognitive training with specific cognitive-motor games. Each training session lasts about 30 to 40 minutes.
  Interventions: Behavioral: Active@Home exergame training
- Control group (No Intervention): Participants of the control group go on with their usual daily life. After post-measurements, they get the Active@Home exergame to use the training system at home. They don't have to follow a specific training plan.

INTERVENTIONS:
Behavioral: Active@Home exergame training — The Active@Home exergame is a multicomponent, motor-cognitive training for fall prevention in elderly adults. It mainly consists of three components; strength training, balance training and cognitive training. For strength training, Tai Chi-based movements are included. For balance training, dancing is included in the Active@Home exergame. Moreover, the Active@Home exergame explicitly targets specific attentional and executive functions. The Active@Home system set up is easy and consists of an HDMI dongle (to run the application) which must be plugged into the TV and four wearable sensors (to measure the movements).
  Arms: Intervention group

SUMMARY:
This study investigates the effects of an exergame training including strength, balance, and cognitive training components on motor functions, cognition and brain structure of older adults. The primary objective is to determine the effects of the home-based multicomponent exergame training on motor and cognitive functions of older adults compared to a usual care waitlist control group. To understand the underlying mechanisms, the secondary objective is to assess the effect of the exergame training on neuronal level (brain structure). The study design is a randomized controlled trial including 40 healthy (self-reported), independently living older adults aged 65 years and older. The intervention period lasts for 16-18 weeks (no longer than two weeks of break/holiday allowed) with three training sessions per week each lasting about 40 minutes.

DETAILED DESCRIPTION:
Age-associated degenerative changes cause gait impairments and a higher risk of falls in elderly. Falls are a leading cause for injuries, reduced mobility, independence and general well-being. Most of the investigator's daily life activities, including walking, are tasks which require not only motor but also cognitive functions. Therefore, also in fall prevention, there is a need for combined motor-cognitive interventions. Exergames - games which require physical activity and movement to play the game - are a promising option for motivating and engaging motor-cognitive training, especially in combination with newly available technologies. In an international project of the Ambient Assisted Living Association (AAL), a new exergame (Active@Home) was developed which ultimately aims for fall prevention in elderly and incorporates theoretical background from movement sciences, neuropsychology, cognitive sciences, and arts of game design.

During aging, age-related changes are evident not only in sensory, motor and cognitive functions but also on (underlying) neuronal level: The aging brain is associated with neurostructural changes and functional changes in neuronal activity pattern. Especially the (pre)frontal lobe and medial temporal lobe (Hippocampus) are vulnerable to age-related degeneration. However, also in higher age, experience-based neuroplasticity can be observed; the adult brain possesses the ability to alter cortical functions and structures in response to stimulation or training. Evidence shows that experience-dependent neural plasticity can be enhanced by both, physical and cognitive exercise. The question arises how a combination of both - combined motor-cognitive training - influences neuroplasticity in the aging brain. Exergame training has been shown to improve motor as well as cognitive functions. To understand the underlying mechanisms of these training effects, the impact on the level of neuronal activity and brain structure has to be studied.

The primary objective of this study is to determine the effects of a home-based multicomponent exergame training on motor and cognitive functions of older adults compared to a usual care waitlist control group.

To understand the underlying mechanisms, the secondary objective is to assess the effect of the exergame training on neuronal level (brain structure).

The Active@Home exergame is a multicomponent, motor-cognitive training for fall prevention in elderly adults. It mainly consists of three components; strength training, balance training and cognitive training. For strength training, Tai Chi-based movements are included as Tai Chi is mainly performed in a semi-squat posture that places a large load on the muscles of the lower extremities. For balance training, dancing is included in the Active@Home exergame as the execution of rapid and well-directed steps has been shown to be effective in preventing falls. Both, Tai Chi and dancing, are 'holistic' physical activities requiring motor functions, cognition and mental involvement. Moreover, the Active@Home exergame explicitly targets specific attentional and executive functions (selective attention, divided attention, inhibition/interference control, mental flexibility, working memory) which are important for walking and safe gait. To maximize benefits for participants, the Active@Home exergame implements some basic general training principles; providing feedback, optimal load of task demands, progression of difficulty and high variability. The Active@Home system set up is easy and consists of an HDMI dongle (to run the application) which must be plugged into the TV and four wearable sensors (to measure the movements).

All interested participants will be screened for eligibility for the study (cognitive screening with MMSE, health screening with questionnaire). Then the eligible participants are randomly allocated to either the intervention group or the waitlist control group. At the first appointment (T1), pre-measurements are conducted (motor and cognitive functions, MRI scans) with all participants. The participants of the intervention group will be equipped with the Active@Home exergame kit and instructed how to set up and use the system at home. The intervention period lasts for 16-18 weeks (no longer than two weeks of break/holiday allowed) with three training sessions per week each lasting about 40 minutes. All participants have to fill in an activity protocol during the whole intervention period. After completing all training sessions (in the intervention group), post-measurements are conducted at T2 with all participants. Measurements will take place at the CERENEO (Swiss clinic and research institute at Vitznau, Lucerne). Participants of the waitlist control group are instructed to continue their usual daily business and activities during the study period. After the post-measurements, they will get the Active@Home exergame for their personal use at home (for several months).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years
* Living independently
* Healthy by self-report
* Able to stand unsupported on feet for at least 10-15 minutes
* Written informed consent signed by the participant
* Not participating in a guided existing physical or cognitive training program
* Possess a TV screen with HDMI connection and some space in front of the screen

Exclusion Criteria:

* Cognitive impairments (Mini Mental State Examination, MMSE ≤ 23)
* Severe health problems (e.g. recent cardiac infarction, uncontrolled diabetes or uncontrolled hypertension)
* Orthopaedic disease leading to mobility impairments (that prevent to stand unsupported on feet for at least 10-15 minutes)
* Neurological disease (e.g. history of stroke or epilepsy, Parkinson disease)
* Alzheimer disease or other forms of dementia
* Acute severe illness
* Rapidly progressive or terminal illness
* Intake of any psychoactive substances (neuroleptics, antidepressants etc.) with an influence on neuroplasticity
* Active participation in a guided strength-balance-aerobic endurance or cognitive training program
* Contraindication for MRI: Any metallic parts within the body, metallic or electronic implants (e.g. heart pacemaker, brain pacemaker, cochlear implants), shunts, stents, protheses, ferromagnetic remnants within the body, strong claustrophobia

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 37 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-04-18 (Actual); Study Completion 2019-04-18 (Actual)

PRIMARY OUTCOMES:
Change in gait speed | Assessment takes place at pre- and post-measurement within two weeks before and after the intervention. Pre- and post-measurement changes are calculated. The gait analysis lasts 5 minutes.
  Gait analysis is conducted under single- and dual-task condition and temporal-spatial gait parameters (gait speed, step length, toe clearance) are measured. Gait analysis is conducted with the Physilog. Gait speed is measured in m/s.
Change in balance | Assessment takes place at pre- and post-measurement within two weeks before and after the intervention. Pre- and post-measurement changes are calculated. The balance test lasts 3 minutes.
  To assess balance, the balance test of the Short Physical Performance Battery (SPPB) is used resulting an a total score of 4 points for the balance tasks (e.g. tandem stance, semit tandem stance, single leg stance). A higher score means a better balance performance.
Change in lower body strength | Assessment takes place at pre- and post-measurement within two weeks before and after the intervention. Pre- and post-measurement changes are calculated. The lower body strength test lasts 1 minute.
  Lower body strength is measured by the 30 Seconds Chair Rises Test of the Senior Fitness Test (SFT) resulting in a number of chair rises participants can perform in 30 seconds.
Change in aerobic endurance | Assessment takes place at pre- and post-measurement within two weeks before and after the intervention. Pre- and post-measurement changes are calculated. The aerobic endurance test lasts 3 minutes.
  Aerobic endurance is assessed by the 2 Minutes Stepping Test of the Senior Fitness Test (SFT) resulting in a number of steps done by the participants in 2 minutes.
Change in step length | Assessment takes place at pre- and post-measurement within two weeks before and after the intervention. Pre- and post-measurement changes are calculated. The gait analysis lasts 5 minutes.
  Gait analysis is conducted under single- and dual-task condition and temporal-spatial gait parameters (gait speed, step length, toe clearance) are measured. Gait analysis is conducted with the Physilog. Step length is measured in m.
Change in minimal toe clearance | Assessment takes place at pre- and post-measurement within two weeks before and after the intervention. Pre- and post-measurement changes are calculated. The gait analysis lasts 5 minutes.
  Gait analysis is conducted under single- and dual-task condition and temporal-spatial gait parameters (gait speed, step length, toe clearance) are measured. Gait analysis is conducted with the Physilog. Minimal toe clearance is measured in cm. Smaller values are related to higher risk of tripping and falling.
Change in mental flexibility | Assessment takes place at pre- and post-measurement within two weeks before and after the intervention. Pre- and post-measurement changes are calculated. The TMT lasts 5 minutes.
  To assess mental flexibility (a part of executive functions), the Trail Making Test (TMT) is used pre- and post-intervention. This paper-pencil-test is resulting in a time value in seconds. Less time needed to conducted the test is related to better performance.
Change in interference control | Assessment takes place at pre- and post-measurement within two weeks before and after the intervention. Pre- and post-measurement changes are calculated. The VST lasts 5 minutes.
  To assess interference control (a part of executive functions), the Victoria Stroop Test (VST) is used pre- and post-intervention. The result is a time value measured in seconds, furthermore, errors are counted. Less time and less errors is related to better performance.
Change in memory functions | Assessment takes place at pre- and post-measurement within two weeks before and after the intervention. Pre- and post-measurement changes are calculated. The WMS-R lasts 5 minutes.
  To assess memory functions, the Wechsler-Memory-Sclae-Revised (WMS-R) is used pre- and post-intervention. The test is resulting in a point score. The maximal point score is 12 points, the minimal point score is 0. Higher scores are related to better performance.

SECONDARY OUTCOMES:
Change in grey matter brain structure | Assessment takes place at pre- and post-measurement within two weeks before and after the intervention. Pre- and post-measurement changes are calculated. The T1-weighted sequence lasts 5 minutes.
  Grey matter brain structure is assessed by structural MRI scan with T1-weighted sequence. The focus of the analysis will be on (pre)frontal structures, the hippocampus and the cerebellum.
Change in white matter brain structure | Assessment takes place at pre- and post-measurement within two weeks before and after the intervention. Pre- and post-measurement changes are calculated. The T2-weighted sequences last 10 minutes.
  White matter brain structure is assessed by structural MRI scan with T2-weighted sequence. The focus is on white matter hyper intensities in the whole brain.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Human Movement Sciences and Sport, ETH Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided